CLINICAL TRIAL: NCT04235478
Title: The Evaluation of Effect of the Cervical İnterlaminar Epidural Steroid İnjection on Quality of Life, Neuropathic Pain and Disability in Patients With Cervical Radiculopathy
Brief Title: Effect of the Cervical Interlaminar Epidural Steroid Injection on Quality of Life, Pain and Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/119
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-01

CONDITIONS: Cervical Disc Herniation; Pain, Neuropathic
Keywords: cervical disc herniation; epidural injection; radicular pain; neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Sodium Chloride; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical interlaminar epidural steroid injecion (Experimental): Floroscopy-guided cervical interlaminar epidural steroid injecion will be applied to the patients with cervical radiculopathy related neck and arm pain
  Interventions: Drug: Combination Product: triamcinolone and saline

INTERVENTIONS:
Drug: Combination Product: triamcinolone and saline — a mixture of 3 mL 0.09%saline and 2 mL 80 mg triamcinolone (kenacort-a)
  Other Names: kenacort-a

SUMMARY:
To evaluate the effect of cervical interlaminar epidural steroid injections on the neuropathic pain, quality of life and disability patients with cervical radiculopathy. After the clinical and MRG evaluations of patients with neck and arm pain, injection was given to eligible patients.

Patients undergone the procedure were evaluated before and after injection for neuropathic pain, quality of life and disability.

DETAILED DESCRIPTION:
Neck and arm pain related to cervical radiculopathy is the second indication for epidural steroid injections after lumbar radiculopathy in the many a pain clinic. In this procedure corticosteroids and local anesthetics were given to the epidural space with fluoroscopy-guided special techniques. The underlying mechanism of action of these epidurally administered medications is not clear and ıt is believed to be due to anti-inflammatory properties of corticosteroids. In addition local anesthetics is thought to be as effective as corticosteroids in spinal pain of various origin. So far, many studies have shown the efficacy of these injections in acute/chronic pain of cervical radiculopathy. Although mixed pain is seen in most of patients, the relationship between pain pattern and treatment response is unclear. This study aims to evaluate the treatment responses of the patients who were diagnosed with neuropathic pain and the patients who weren't by means of LANSS. It is also intended to serach whether the presence of neuropathic pain will help to predict the treatment response or not. In this regard, the patients were evaluated with LANSS, SF-12 and neck pain and disability scale before the procedure. Categorized as the patients with neuropathic pain and the patients without, their treatment responses were compared.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain and / or unilateral arm pain for at least 3 months
* Inadequate response to conservative treatment methods
* Visual analog scale>5
* Treatment of neuropathic pain:

Patients who received adequate treatment for a sufficient period of time (Gabapentine ( ≥4 wk ve ≥ 1200 mg) or Pregabaline ( ≥4 wk ve ≥ 300mg )) and did not respond adequately

Exclusion Criteria:

* Cervical epidural injection history applied in the last 3 months
* Presence of systemic and / or local infection
* Bleeding diathesis
* Pregnancy
* Presence of a history of allergy to contrast agent and local anesthetic agent
* Systemic inflammatory disease ( rheumatoid arthritis, SLE..)
* Presence of malignancy
* Presence of polyneuropathy, multiple sclerosis or demyelinating nervous system diseases
* Patients with a history of surgical operations for cervical disc hernia and / or spinal stenosis
* Patients with myelomalacia due to spinal cord compression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain relief | before treatment(T0)
  Pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable) The primary outcome measure is reduction in initial VAS , treatment success was considered a 50% or more reduction in VAS point
Pain relief | 1th month after procedure (T1)
  Pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable) The primary outcome measure is reduction in initial VAS , treatment success was considered a 50% or more reduction in VAS point
Pain relief | 3th month after procedure (T2)
  Pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable) The primary outcome measure is reduction in initial VAS , treatment success was considered a 50% or more reduction in VAS point
Pain relief | 6th month after procedure (T3)
  Pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable) The primary outcome measure is reduction in initial VAS , treatment success was considered a 50% or more reduction in VAS point
Pain classification-The leeds assesment of neuropathic signs&symptoms (LANSS) | before treatment(T0)
  LANSS is an assessment tool that used to analyze and classify pain. The scale comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.According to various research reports, these LANSS tests correctly classified the patients as suffering from nociceptive and neuropathic pain, in four out of every five patients experiencing chronic pain. The validity and reliability of the questionnaire in Turkish were conducted by Yucel et al.
Pain classification-The leeds assesment of neuropathic signs&symptoms (LANSS) | 1th month after procedure (T1)
  LANSS is an assessment tool that used to analyze and classify pain. The scale comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.According to various research reports, these LANSS tests correctly classified the patients as suffering from nociceptive and neuropathic pain, in four out of every five patients experiencing chronic pain. The validity and reliability of the questionnaire in Turkish were conducted by Yucel et al.
Pain classification-The leeds assesment of neuropathic signs&symptoms (LANSS) | 3th month after procedure (T2)
  LANSS is an assessment tool that used to analyze and classify pain. The scale comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.According to various research reports, these LANSS tests correctly classified the patients as suffering from nociceptive and neuropathic pain, in four out of every five patients experiencing chronic pain. The validity and reliability of the questionnaire in Turkish were conducted by Yucel et al.
Pain classification-The leeds assesment of neuropathic signs&symptoms (LANSS) | 6th month after procedure (T3)
  LANSS is an assessment tool that used to analyze and classify pain. The scale comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.According to various research reports, these LANSS tests correctly classified the patients as suffering from nociceptive and neuropathic pain, in four out of every five patients experiencing chronic pain. The validity and reliability of the questionnaire in Turkish were conducted by Yucel et al.

SECONDARY OUTCOMES:
Quality of life-Short form-12 | before treatment(T0)
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. The SF-12 consists of a subset of 12 items from the SF-36. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).SF-12 scales and summary measures are scored so that a higher score indicates a better health state.
Quality of life-Short form-12 | 1th month after procedure (T1)
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. The SF-12 consists of a subset of 12 items from the SF-36. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).SF-12 scales and summary measures are scored so that a higher score indicates a better health state.
Quality of life-Short form-12 | 3th month after procedure (T2)
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. The SF-12 consists of a subset of 12 items from the SF-36. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).SF-12 scales and summary measures are scored so that a higher score indicates a better health state.
Quality of life-Short form-12 | 6th month after procedure (T3)
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. The SF-12 consists of a subset of 12 items from the SF-36. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).SF-12 scales and summary measures are scored so that a higher score indicates a better health state.
Disability-Neck pain and disability scale (NPAD) | before treatment(T0)
  The Neck Pain and Disability scale (NPAD) is a composite index including 20 items which measure the intensity of neck pain and related disability. Patients respond to each item by marking along a 10cm visual analog scale (VAS). Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)).a High scores are associated with increased disability.
Disability-Neck pain and disability scale (NPAD) | 1th month after procedure (T1)
  The Neck Pain and Disability scale (NPAD) is a composite index including 20 items which measure the intensity of neck pain and related disability. Patients respond to each item by marking along a 10cm visual analog scale (VAS). Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)).a High scores are associated with increased disability.
Disability-Neck pain and disability scale (NPAD) | 3th month after procedure (T2)
  The Neck Pain and Disability scale (NPAD) is a composite index including 20 items which measure the intensity of neck pain and related disability. Patients respond to each item by marking along a 10cm visual analog scale (VAS). Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)).a High scores are associated with increased disability.
Disability-Neck pain and disability scale (NPAD) | 6th month after procedure (T3)
  The Neck Pain and Disability scale (NPAD) is a composite index including 20 items which measure the intensity of neck pain and related disability. Patients respond to each item by marking along a 10cm visual analog scale (VAS). Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)).a High scores are associated with increased disability.
cervical range of motion (ROM) will be evaluated with a goniometer | before treatment(T0)
  cervical range of motion (ROM) will be evaluated with a goniometer all directions
cervical range of motion (ROM) will be evaluated with a goniometer | 1th month after procedure (T1)
  cervical range of motion (ROM) will be evaluated with a goniometer all directions
cervical range of motion (ROM) will be evaluated with a goniometer | 3th month after procedure (T2)
  cervical range of motion (ROM) will be evaluated with a goniometer all directions
cervical range of motion (ROM) will be evaluated with a goniometer | 6th month after procedure (T3)
  cervical range of motion (ROM) will be evaluated with a goniometer all directions
upper extremity motor exam | before treatment(T0)
  Muscle strength is tested from the proximal to the distal part of the upper extremity so that all segmental levels for the extremity will be tested according to the a scale of 0/5 to 5/5. İn addition upper extremity deep tendon relfex will also evalutaed
upper extremity motor exam | 1th month after procedure (T1)
  Muscle strength is tested from the proximal to the distal part of the upper extremity so that all segmental levels for the extremity will be tested according to the a scale of 0/5 to 5/5. İn addition upper extremity deep tendon relfex will also evalutaed
upper extremity motor exam | 3th month after procedure (T2)
  Muscle strength is tested from the proximal to the distal part of the upper extremity so that all segmental levels for the extremity will be tested according to the a scale of 0/5 to 5/5. İn addition upper extremity deep tendon relfex will also evalutaed
upper extremity motor exam | 6th month after procedure (T3)
  Muscle strength is tested from the proximal to the distal part of the upper extremity so that all segmental levels for the extremity will be tested according to the a scale of 0/5 to 5/5. İn addition upper extremity deep tendon relfex will also evalutaed

CONTACTS AND LOCATIONS:
Overall Officials: Savaş ŞENCAN, Asst. Prof, Principal Investigator — Marmara University
Locations (1):
- Feyza Nur YUCEL, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner-Bowker D., Hogue S.J. (2014) Short Form 12 Health Survey (SF-12). In: Michalos A.C. (eds) Encyclopedia of Quality of Life and Well-Being Research. Springer, Dordrecht
- [Result] Manchikanti L, Nampiaparampil DE, Candido KD, Bakshi S, Grider JS, Falco FJ, Sehgal N, Hirsch JA. Do cervical epidural injections provide long-term relief in neck and upper extremity pain? A systematic review. Pain Physician. 2015 Jan-Feb;18(1):39-60. PMID 25675059
- [Result] Yucel A, Senocak M, Kocasoy Orhan E, Cimen A, Ertas M. Results of the Leeds assessment of neuropathic symptoms and signs pain scale in Turkey: a validation study. J Pain. 2004 Oct;5(8):427-32. doi: 10.1016/j.jpain.2004.07.001. PMID 15501424
- [Derived] Sanal-Toprak C, Ozturk EC, Yucel FN, Sencan S, Gunduz OH. Does the presence of neuropathic pain affect the outcomes of the interlaminar epidural steroid injection for cervical disc herniation?: A prospective clinical study. Medicine (Baltimore). 2021 Mar 5;100(9):e25012. doi: 10.1097/MD.0000000000025012. PMID 33655971